CLINICAL TRIAL: NCT07388771
Title: A Study on Multimodal Data Prediction of Outcome to Neoadjuvant Therapy in NSCLC
Brief Title: Prediction of Outcome to Neoadjuvant Therapy in Non-small Cell Lung Cancer（NSCLC）
Status: Recruiting | Type: Observational
Sponsor: Qian Chu (Other)
Responsible Party: Sponsor-Investigator, Qian Chu, Director of the Thoracic Oncology Department, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202512147
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: NSCLC; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Preoperative pathological biopsy puncture specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC with neoadjuvant therapy but without surgery
- NSCLC with neoadjuvant therapy and surgery

SUMMARY:
This observational study aims to construct and validate the performance of a multimodal predictive model in forecasting the outcomes of neoadjuvant therapy in patients with NSCLC.

The core research question is: Can a multi-model approach predict outcomes of neoadjuvant therapy for non-small cell lung cancer and provide clinical recommendations?

ELIGIBILITY:
Inclusion Criteria:

1. pathologically diagnosed non-small cell lung cancer
2. The treatment plan is：receiving neoadjuvant chemo-immunotherapy during the study period, followed by surgical resection

Exclusion Criteria:

1. recurrent or metastatic lung cancer;
2. patients with other primary tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients suitable for neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
pathologic response | Perioperative

SECONDARY OUTCOMES:
EFS | One year after the treatment ended
  event free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Due to patient and hospital ethical requirements, this project does not currently meet the criteria for Individual Patient Data (IPD).